CLINICAL TRIAL: NCT03535389
Title: Morphological and Biomechanical Analysis of Knee 4DCT in Femoropatellar Instability
Brief Title: Morphological and Biomechanical Analysis of Knee Four Dimensional CT (4DCT) in Femoropatellar Instability
Acronym: EDYG
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 2018-A00450-55
Record Dates: First submitted 2018-05-14; First posted 2018-05-24 (Actual); Last update posted 2019-06-10 (Actual); Status verified 2019-06

CONDITIONS: 4DCT, Knee, Femoropatellar Instability

STUDY DESIGN:
Intervention Model Description: Case-control study, cross-sectional, monocentric, with prospective recruitment.
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pathologic group (Experimental): Patients addressed to our imaging department for the realization of a knee scanner as part of routine care and presenting clinical PFI syndrome (Patellofemoral instability diagnosis based on physical examination, history and Kujala score)
  Interventions: Diagnostic Test: Knee 4DCT
- Control group (Active Comparator): Patients addressed to our imaging department for osteo-articular pathologies other than patellofemoral instability (non-fracture trauma, vascular pathologies, degenerative or soft tissues).
  * Does not have any clinical PFI syndrome
  * Matched (1: 1 ratio) to PFI patients by age (+/- 40 years) and sex
  Interventions: Diagnostic Test: Knee 4DCT

INTERVENTIONS:
Diagnostic Test: Knee 4DCT — Dynamic knee 4DCT

SUMMARY:
To compare the radiological parameters measured by dynamic four dimensional CT (4DCT) in the analysis of patellofemoral involvement of subjects (amplitude of patellofemoral tilt angle variations, coefficient of variation of the same angle, distance of lateral displacement of the patella ) in patients with patellofemoral clinical syndrome to those free of this syndrome (= control group).

It is expected that the amplitude of patellofemoral tilt angle changes, its coefficient of variation, and the patella lateral displacement distance differ between the 2 groups compared. This result would clarify the potential value of dynamic 4D CT in the diagnosis of PFI

DETAILED DESCRIPTION:
Patellofemoral instability (PFI) is frequent, causing chronic knee pain, functional impotence or disability because it is associated with the development of early patellofemoral osteoarthritis. PFI are classically classified into three types: anterior pain syndrome (SR, without structural abnormality), potential patellar instability (with structural anomaly favoring, but no history of patellar dislocation) and objective patellar instability (with structural abnormality and history of patellar dislocation). Diagnosis of the disease outside objective patellar instability is difficult at present, and objective criteria are lacking to determine management and evaluate the rehabilitation program of these patients.

Radiographic assessment of the knee is the diagnostic method of reference to objectify patellar patellofemoral instability and to look for contributing factors including signs of trochlear dysplasia, and remains the initial method of exploration of a patellar syndrome. Static imaging reveals signs of objective instability (patellar luxation, fracture stigmas) or favorite factors (trochlear dysplasia, increased distance of anterior tibial tuberosity / trochlear throat).

Nevertheless, some important elements in the pathophysiology of patellofemoral instability such as patellar tilt and lateral displacement of the patella are essentially dynamic and vary according to the degree of flexion-extension of the knee. Our hypothesis is that the variation of these parameters during the movements could make it possible to improve the diagnosis of patellar instabilities without favoring structural anomaly and the follow-up of the patients who benefit from a patellofemoral reeducation program.

Some authors propose functional MRI of the knee with static acquisitions during different movements. Nevertheless, no validated technique allows the study of biodynamic anomalies in real time. The dynamic knee scanner is not very radiating and the knee is not very radio-sensitive. This technique could therefore represent an interesting alternative allowing dynamic analysis of patellar displacements during knee flexion and patellar engagement. Finally, new methods of post-processing CT images based on registration and automatic segmentation of bone structures are available for clinical application. This type of tool allows a semi-automatic quantification of patellar displacements that could provide objective evaluation criteria for patients with patellofemoral instability. In 2016, a Swedish team published a study on the feasibility of five patients performing a quantitative semi-automatic dynamic scanner analysis of patellofemoral flexion-extension joint movement. This shows the value of evaluating this method in a larger population with a control group

Main objective: To compare the radiological parameters measured by dynamic 4D CT in the analysis of patellofemoral involvement of subjects (amplitude of patellofemoral tilt angle variations, coefficient of variation of the same angle, distance of lateral displacement of the patella ) in patients with patellofemoral clinical syndrome (= Cas group) to those free of this syndrome (= control group).

It is expected that the amplitude of patellofemoral tilt angle changes, its coefficient of variation, and the patella lateral displacement distance differ between the 2 groups compared. This result would clarify the potential value of dynamic 4D CT in the diagnosis of PFI.

Secondary objectives:

1. compare, in the pathologic group, the radiological parameters measured by 4D dynamic CT (coefficient of variation, amplitude of the patellofemoral tilt angle and distance of patella lateral displacement) according to the type of patellofemoral instability ( anterior pain syndrome, potential patellar femoro instability and "objective" femoro-patellar instability) obtained by conventional imaging (static CT).
2. To estimate the interobserver reproducibility of the radiological parameters measured by 4D dynamic CT during image post-treatment in all patients (measurement of patellofemoral angle of flap angle and distance of patella lateral displacement)

ELIGIBILITY:
Inclusion Criteria:

* Patient between 18 and 60 years old
* giving consent
* Mandatory affiliation to a social security scheme

  * patients with clinical symptoms of femoropatellar instability addressed for a knee CT scan

Pathologic group:

* Consultant at our institution's imaging department for the realization of a knee scanner as part of routine care.
* Presenting clinical PFI syndrome (Patellofemoral instability diagnosis based on physical examination, history and Kujala score)

Control group:

* Consultant at our institution's imaging department for osteo-articular pathologies other than PFI (non-fracture trauma, vascular pathologies, degenerative or soft tissues).
* Does not have any clinical PFI syndrome
* Matched (1: 1 ratio) to PFI patients by age (+/- 40 years) and sex

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-06 (Estimated); Primary Completion 2019-06 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
• Amplitude (in °) of patellofemoral angle | 2 years
  Amplitude of changes in patellofemoral angle measured by 4D dynamic CT in the analysis of patellofemoral involvement in the 2 subgroups (Cases and controls);
Coefficient of variation of patellofemoral tilt angle | 2 years
  (standard deviation / mean)
Distance of lateral displacement of the patella (in mm) | 2 years

SECONDARY OUTCOMES:
Amplitude (in °) of changes in patellofemoral angle, coefficient of variation of patellofemoral tilt angle and distance of patella lateral displacement (in mm) | 2 years
Intra-class correlation coefficient | 2 years

IPD SHARING:
Plan to Share IPD: Undecided